CLINICAL TRIAL: NCT01037348
Title: A Phase II, Open-label, Multicentre, 12 Month Study to Evaluate the Efficacy and Safety of Ranibizumab (0.5mg) in Patients With Choroidal Neovascularisation Secondary to Pathological Myopia (PM)
Brief Title: Ranibizumab for the Treatment of Choroidal Neovascularisation (CNV) Secondary to Pathological Myopia (PM): an Individualized Regimen
Acronym: REPAIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002AGB10; 2009-014854-14 (EudraCT Number)
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Choroidal Neovascularisation
Keywords: Choroidal Neovascularisation; Pathological Myopia
MeSH Terms: conditions — Choroidal Neovascularization; Myopia, Degenerative | interventions — Ranibizumab

ARMS (1):
- ranibizumab 0.5mg (Experimental)
  Interventions: Drug: ranibizumab 0.5mg

INTERVENTIONS:
Drug: ranibizumab 0.5mg

SUMMARY:
This study is designed to provide efficacy and safety data in patients with choroidal neovascularisation (CNV) secondary to myopia using an individualized as-needed (PRN) dosing schedule. Eligible patients who have provided written agreement to take part in the study will receive an intravitreal (into the study eye) injection of ranibizumab 0.5mg. Following eye examinations and tests at monthly clinic visits, the study doctor will repeat the injections on a monthly basis as required for an additional 11 months, in accordance with specified retreatment criteria.

Patients will be in the study for approximately 12 months and will visit the hospital clinic 14 times over that period. The main assessments will include visual acuity tests, eye examinations, optical coherence tomography (OCT) to assess retinal thickness, fundus photography and fluorescein angiography (FA), measurement of intraocular pressure, blood pressure and pulse measurements and completion of health-related questionnaires'.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients of any race, aged 18 years or older
* Diagnosis of active primary or recurrent subfoveal or juxtafoveal CNV secondary to PM
* Diagnosis of high myopia of at least -6 dioptres in the study eye spherical equivalent. For subjects who have undergone prior refractive or cataract surgery in the study eye, the preoperative refractive error in the study eye must have been at least -6 dioptres
* Patients who have a BCVA score between 78 and 24 letters in the study eye using Early Treatment Diabetic Retinopathy Study (ETDRS)-like grading charts (approximately 6/9 - 6/96 Snellen equivalent)
* Patients must give fully informed consent and be willing and able to comply with all study procedures

Exclusion Criteria:

* History of any surgical intervention in the study eye within two months preceding screening
* Previous macular laser photocoagulation, treatment with intravitreal steroids, verteporfin with photodynamic therapy (Visudyne®) or anti-VEGF agents ranibizumab, bevacizumab or pegaptanib sodium (Macugen®) in the study eye
* Previous treatment with intravenously administered bevacizumab (Avastin®)
* Prior treatment in the study eye with external-beam radiation therapy, vitrectomy, or transpupillary thermotherapy
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
* History of allergic reaction to fluorescein
* Concurrent use of systemic anti-VEGF agents

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The difference from baseline in mean Best Corrected Visual Acuity (BCVA) | 12 months

SECONDARY OUTCOMES:
Mean change in BCVA from baseline | 6 months
Mean change in Central retinal Thickness (CRT) from baseline | 6 and 12 months
Percentage of patients gaining ≥ 15 letters | 12 months
Change in lesion size and morphology from baseline | 6 and 12 months
Time to the first retreatment and the total number of treatments | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United Kingdom (11):
  - Novartis Investigative Site, Bristol
  - Novartis Investigational Site, City of London
  - Novartis Investigative Site, City of London
  - Novartis Investigative Site, Frimley
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Torquay
  - Novartis Investigative Site, Wolverhampton
  - Novartis Investigative Site, York

REFERENCES:
- [Derived] Tufail A, Narendran N, Patel PJ, Sivaprasad S, Amoaku W, Browning AC, Osoba O, Gale R, George S, Lotery AJ, Majid M, McKibbin M, Menon G, Andrews C, Brittain C, Osborne A, Yang Y. Ranibizumab in myopic choroidal neovascularization: the 12-month results from the REPAIR study. Ophthalmology. 2013 Sep;120(9):1944-5.e1. doi: 10.1016/j.ophtha.2013.06.010. No abstract available. PMID 24001532